CLINICAL TRIAL: NCT04930666
Title: The Development and Pilot Testing of a Brief Shared Decision-Making Intervention to Improve Palliative Care Outcomes for Adults With Advanced Lung Disease
Brief Title: BREATHE ALD: A Shared Decision-Making Intervention for Adults With Advanced Lung Disease
Acronym: BREATHE-ALD
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maureen George, Professor of Nursing at CUIMC, Columbia University
Other Study IDs: AAAT2217; P20NR018072 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial
Keywords: Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: BRief intervention to Enhance Adherence to Treatment and HEalth advice in Advanced Lung Disease — BREATHE-ALD utilizes the patient's nurse practitioner (NP) to deliver a brief intervention using motivational interviewing and shared decision making, in a one-time 9-minute intervention. The NP will follow a 4-step script tailored to specific ALD self-management discussed during the most recent visit with the patient's pulmonologist. Step 1: Raise the subject (1½ minute). Step 2: Provide feedback (1½ minutes). Step 3: Enhance engagement (3 minutes). Step 4: Shared decision-making (3 minutes).
  Other Names: BREATHE-ALD

SUMMARY:
This study aims to:

1. Develop the BREATHE-ALD intervention for adults with Advanced Lung Disease, multiple chronic conditions, and palliative care needs and their caregivers using interviews with 10 advanced lung disease (ALD) adults and their caregivers
2. To evaluate the feasibility and acceptability of intervention procedures; and
3. To explore intervention effects on ALD outcomes

DETAILED DESCRIPTION:
This study addresses the important problem of adults with symptomatic advanced lung disease (ALD) who are at high risk for poor outcomes. Palliative care (PCare) improves the quality of life of individuals and their caregivers through the prevention and relief of suffering by identifying, assessing and treating the physical, psychosocial and spiritual problems associated with life-threatening illness. However, pulmonary clinicians rarely refer adults with ALD to PCare because of time demands, a lack of confidence in PCare and the perceived threat PCare poses to the relationship they have established with the ALD adult. Therefore, we are developing BREATHE-ALD (BRief intervention to Enhance Adherence to Treatment and HEalth advice in Advanced Lung Disease [ALD]), a novel shared decision-making (SDM) intervention to improve outcomes for adults with ALD.

The study includes two phases: (1) a development phase to develop BREATHE-ALD using interviews with 10 ALD adults and their caregivers with expert review to adapt BREATHE, and (2) a pilot validation phase conducting a pilot trial in which 10 adults with ALD receive BREATHE-ALD. We will follow adults with ALD for 3 months post-intervention to assess the impact of BREATHE-ALD on self-management and patient outcomes.

ELIGIBILITY:
Pre-trial

Inclusion Criteria:

* Patient participants with symptomatic advanced lung disease (ALD) followed at Weill Cornell Medicine (WCM).
* Caregiver participants who care for adults with symptomatic ALD followed at Weill Cornell Medicine.

Exclusion Criteria:

* Patients that have serious mental health conditions that preclude completion of study procedures or confound analyses.
* Caregivers that have serious mental health conditions that preclude completion of study procedures or confound analyses.

Trial

Inclusion Criteria:

* Patient participants with symptomatic advanced lung disease (ALD) followed at Weill Cornell Medicine (WCM).
* Nurse practitioner must manage a panel of adult ALD patients.

Exclusion Criteria:

* Patients that have serious mental health conditions that preclude completion of study procedures or confound analyses.
* Patients anticipated to have less than 3-month survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and caregivers of patients followed for advanced lung disease at Weill Cornell Medicine. Nurse practitioner who manages ALD patients at Weill Cornell Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Number of qualitative interviews completed in the development phase | Up to 6 months
  Qualitative interviews will be conducted with adults with advanced lung disease and their caregivers to understand their experiences managing ALD using semi-structured in-depth individual interviews. The information collected will aid the design of BREATHE-ALD and the implementation of the pilot phase of this study.
Ratio of participants who completed the intervention to the number of participants consented | Up to 3 months post-intervention
  To determine the level of retention, the ratio of participants who completed the intervention to the number of participants consented will be measured.
Mean mMRC (Modified Medical Research Council) Dyspnea Scale | Up to 3 months post-intervention
  The mMRC (Modified Medical Research Council) Dyspnea Scale measures the effect of breathlessness when performing daily activities. The mMRC breathlessness scale comprises ﬁve statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5).

SECONDARY OUTCOMES:
Mean St. George's Respiratory Questionnaire | Baseline, 1 month, 2 months, and 3 months (post-intervention)
  The St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. It is a 50-item questionnaire with two parts, in which part one measures frequency and severity of symptoms while part two measures activities that impact breathlessness. Scores range from 0 to 100, with higher scores indicating more limitations.
Mean PROMIS Pain Intensity - Short Form V10 3a | Baseline, 1 month, 2 months, and 3 months (post-intervention)
  PROMIS Pain Intensity instrument measures how much a person hurts. It is a 3-item instrument that evaluates how much pain the patient has felt in the past seven days. Each question about pain intensity is rated on a five-point scale from had no pain (1) to very severe (5).
Mean PROMIS Fatigue - Short Form 6a | Baseline, 1 month, 2 months, and 3 months (post-intervention)
  PROMIS Fatigue instrument measures how much a person feels tired. It is a 6-10-item questionnaire that evaluates how tired or exhausted the patient has felt in the past seven days. Each question about fatigue is rated on a five-point scale from never (1) to always (5).
Mean Short Form 36 | Baseline, 1 month, 2 months, and 3 months (post-intervention)
  Short Form 36 (SF-36) is a well validated instrument that measures overall health status. It consists of 36 items and has eight sections.; the scores are weighted sums of the questions in each section. Scores range from 0-100. Lower scores = more disability and higher scores = less disability
Mean Shared Decision Making Questionnaire | Baseline (immediately post-intervention)
  The Shared Decision Making (SDM) Questionnaire-9, is a patient reported, 9-item validated instrument that consists of nine statements that measure the decisional process in medical visits from both patients' and physicians' perspectives. Each statement is rated on a six-point scale from "completely disagree" to "completely agree".

CONTACTS AND LOCATIONS:
Overall Officials: Maureen George, PhD, Principal Investigator — Columbia University School of Nursing
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States